CLINICAL TRIAL: NCT06322459
Title: Effect of Football's Sport Education Curriculum as Intervention on Physical Fitness and Learning Attitude Among Junior High School Students in Hebei China
Brief Title: Effect of Sport Education on Physical Fitness and Learning Attitude Among Junior High School Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Junlong Zhang, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Junlong Zhang
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Physical Fitness
Keywords: Football teaching; Physica fitness; Cognitive; Affective

STUDY DESIGN:
Intervention Model Description: Employing a Cluster randomized controlled experiment design, the experimental and control groups were randomly assigned to two different schools. Students participated in the Sport Education Model (experimental group) and traditional teaching (control group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sport Eucation Curriculum (Experimental): The Teaching experiment period of the Sport Education Model was 12 weeks, 40 minutes per lesson which included warm-up (10 minutes), basic content (20 minutes), rest of basic content (5 minutes), and cool-down (5 minutes).
  Interventions: Behavioral: Sport Education Curriculum
- Normal Teaching (Active Comparator): The Teaching experiment period of Normal Teaching was 12 weeks, 40 minutes per lesson which included warm-up (10-min), basic content (20min), rest of basic content (5min), and cool-down (5min). Normal Teaching includes Teacher-directed learning (10 minutes) and Individual practice (10 minutes).
  Interventions: Behavioral: Normal teaching

INTERVENTIONS:
Behavioral: Sport Education Curriculum — The six characteristics of The Sport Education Model include season, affiliation, formal competition, culminating event, Record-keeping, and Festivity. The intensity of the training is increasing in the first 30 minutes, and the intensity is gradually decreasing in the next 10 minutes.
  Arms: Sport Eucation Curriculum
Behavioral: Normal teaching — The intervention content, frequency, and intensity were the same as those in the experimental group, but the type of intervention was different. The most significant difference between the two teaching methods lies in delivering basic content. The Sport Education Model includes Teacher-directed learning (10 minutes) and Team practice (10 minutes); Normal Teaching includes Teacher-directed learning (10 minutes) and Individual practice (10 minutes).
  Arms: Normal Teaching

SUMMARY:
Since the outbreak of COVID-19, students; sports environment and time have been severely compressed, which has had an unprecedented impact on their physical fitness and sports learning attitude. Therefore, it is urgent to adopt an effective teaching mode that aligns with curriculum reform to improve students; physical quality and learning attitude. The Sports Education Model is one of the most popular teaching models in Western developed countries, but the application in China and the related evidence of improving students; physical quality and learning attitude towards sports are relatively scarce. This study compares and analyzes the influence of the Sports Education Model and Traditional Teaching on junior middle school students; physical fitness and learning attitude, aiming to provide theoretical support for improving students; physical fitness and learning attitude and promoting the Sports Education Model in China. Promote the healthy development of junior middle school students.

DETAILED DESCRIPTION:
In the study, the experimental group underwent a 12-week soccer program based on the Sport Education Model instructional intervention designed for this research. In contrast, the control group discussed and studied traditional soccer teaching content for 12 weeks with their teachers. Employing a Cluster randomized controlled experiment design, the experimental and control groups were randomly assigned to two different schools. Students participated in the Sport Education Model (experimental group) and traditional teaching (control group) sessions three times a week, each lasting 40 minutes (totaling 120 minutes per week). Physical fitness tests and responses to the Students' Attitudes Toward Physical Education Scale (SPEA) were conducted for both groups before the start of the first week. After 12 weeks of instruction, both groups were required to undergo physical fitness tests and respond to the Students' Attitudes Toward Physical Education Scale once again.

ELIGIBILITY:
Inclusion Criteria:

The experimental subjects were students from two junior high schools in Haigang District, Qinhuangdao City, Hebei province. Before enrolling subjects, researchers need to inform them of the proposed study and what they need to participate in. After the subject is informed, the subject is allowed to ask questions. The various criteria and requirements for participation in this study were explained during the meeting. The criteria for inclusion of potential participants are as follows:

1. Participants must be enrolled in junior high school and mixed gender.
2. Participants must be in good health and capable of engaging in regular physical education activities.
3. All participants and their parents have provided written informed consent for their involvement in the study.

Exclusion Criteria:

1. Participants failing to complete all tests due to attendance-related issues (25%) or illness during experimental teaching or testing will be excluded.
2. Participants who have already participated in the Sport Education Model will be excluded.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular fitness test | Pretest: before experiment; post-test1: end of 6 weeks; post-test2: end of 12 weeks
  Equipment: Soccer field, cones, tape measure, Yo-Yo test software. Procedure: Warm-up, group athletes, select appropriate mode, shuttle runs between cones with increasing speed, complete each run between beeps, record last completed run, measure total distance in meters (m).
Flexibility test | Pretest: before experiment; post-test1: end of 6 weeks; post-test2: end of 12 weeks
  Equipment: Sit and reach box. Procedure: Participant sits, feet against box, knees extended, bends forward reaching forward with fingertips, measure maximum range without sudden force, knees remain extended, retest if technical issues, measure in centimeters (cm).
Speed test | Pretest: before experiment; post-test1: end of 6 weeks; post-test2: end of 12 weeks
  Equipment: Soccer field, tape measure, timing gates or stopwatch, cones or poles.
  Procedure: Thoroughly warm up, sprint 30 meters twice, record the best time, calculated in seconds (s).

CONTACTS AND LOCATIONS:
Overall Officials: Junlong Zhang, Principal Investigator — University Putra Malaysia
Locations (1):
- The 19th Middle School, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.